CLINICAL TRIAL: NCT01156363
Title: A Single Arm, Open Label Study to Assess the Efficacy, Safety and Tolerability of Once-monthly Administration of Subcutaneous and Intravenous MIRCERA® for the Maintenance of Haemoglobin Levels in Dialysis Patients With Chronic Renal Anaemia
Brief Title: A Study of Monthly Subcutaneous or Intravenous Mircera in Dialysis Patients With Chronic Renal Anaemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22299
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-10

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Dialysis; continuous erythropoietin receptor activator

ARMS (1):
- Single Arm (Experimental)
  Interventions: Procedure: Dialysis; Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Procedure: Dialysis — regular haemodialysis or peritoneal dialysis
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — once monthly, subcutaneously or intravenously, for 32 weeks

SUMMARY:
This open label, single arm study will assess the efficacy for long-term maintenance of haemoglobin levels and the safety and tolerability of methoxy polyethylene glycol-epoetin beta [Mircera] in dialysis patients with chronic renal anaemia. Patients on regular long-term haemodialysis or peritoneal dialysis will receive monthly subcutaneous or intravenous Mircera for 6 months. Target sample size is <200 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* chronic renal anaemia
* haemoglobin 10.0-12.0g/dl at screening
* adequate iron status
* continuous stable ESA (erythropoietic stimulating agent) therapy for >/= 2 months
* regular haemodialysis or regular peritoneal dialysis for >/= 3 months

Exclusion Criteria:

* uncontrolled hypertension
* haemoglobinopathy
* anaemia due to haemolysis
* pure red cell aplasia (PRCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Taiwan (3):
  - Kaohsiung City
  - New Taiepei City
  - Taichung

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Efficacy results are reported separately for each of the 3 centers involved in the study [China Medical University Hospital (CMUH); Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH); and Buddhist Tzu Chi General Hospital (BTCH)] as well as for overall treatment arm, unless otherwise specified.
Groups:
- Mircera: Participants received Mircera (epoetin beta-methoxy polyethylene glycol) 80, 120, 200, or 360 micrograms (mcg) (based on the weekly dose of erythropoiesis stimulating agent [ESA] participant received in the week preceding the switch to Mircera [Week -1]) by intravenous (IV) or subcutaneous (SC) injection once monthly for a total of 32 weeks. Doses were adjusted, if required, based on hemoglobin (Hb) level.
  This arm includes participants enrolled at all 3 centers.
Period: Overall Study
Arm/Group | Mircera
Started | 86
Completed | 64
Not Completed | 22
Not completed — Adverse Event | 6
Not completed — Insufficient Therapeutic Response | 5
Not completed — Failure to Return | 1
Not completed — Refused Treatment | 4
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included participants who had received at least 1 dose of Mircera (Week 0) and for whom data for at least one follow-up variable was available.
Groups:
- Mircera: Participants received Mircera 80, 120, 200, or 360 mcg (based on the weekly dose of ESA participant received in the week preceding the switch to Mircera) by IV or SC injection once monthly for a total of 32 weeks. Doses were adjusted, if required, based on Hb level.
  This arm includes participants enrolled at all 3 centers.
Arm/Group | Mircera
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Average Hemoglobin (Hb) Concentration Within the Target Range
Description: Percentage of participants who maintained the Hb concentration within target range (between 10.0 and 12.0 grams per deciliter [g/dL]) throughout the treatment period were reported.
Time Frame: Weeks 1 to 32
Population: ITT Population.
Measure: Number; unit: percentage of participants
Groups:
- Mircera - CMUH: Participants received Mircera 80, 120, 200, or 360 mcg (based on the weekly dose of ESA participant received in the week preceding the switch to Mircera [Week -1]) by IV or SC injection once monthly for a total of 32 weeks. Doses were adjusted, if required, based on Hb level.
  This arm includes participants enrolled at China Medical University Hospital (CMUH).
- Mircera - KMUH: Participants received Mircera 80, 120, 200, or 360 mcg (based on the weekly dose of ESA participant received in the week preceding the switch to Mircera [Week -1]) by IV or SC injection once monthly for a total of 32 weeks. Doses were adjusted, if required, based on Hb level.
  This arm includes participants enrolled at Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH).
- Mircera - BTCH: Participants received Mircera 80, 120, 200, or 360 mcg (based on the weekly dose of ESA participant received in the week preceding the switch to Mircera [Week -1]) by IV or SC injection once monthly for a total of 32 weeks. Doses were adjusted, if required, based on Hb level.
  This arm includes participants enrolled at Buddhist Tzu Chi General Hospital (BTCH).
- Mircera: Participants received Mircera 80, 120, 200, or 360 mcg (based on the weekly dose of ESA participant received in the week preceding the switch to Mircera [Week -1]) by IV or SC injection once monthly for a total of 32 weeks. Doses were adjusted, if required, based on Hb level.
  This arm includes participants enrolled at all 3 centers.
Arm/Group | Mircera - CMUH | Mircera - KMUH | Mircera - BTCH | Mircera
Number analyzed (Participants) | 35 | 26 | 22 | 83
percentage of participants | 77.1 | 88.5 | 90.9 | 84.3

2. Secondary Outcome: Mean Monthly Hb Values
Description: The baseline (reference) hemoglobin was defined as the average of the three assessments recorded during the screening and baseline visits (Week -2, -1, and 0).
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8
Population: ITT Population. Here, n signifies participants evaluable at specified time-point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Mircera - CMUH: Participants received Mircera 80, 120, 200, or 360 mcg (based on the weekly dose of ESA participant received in the week preceding the switch to Mircera [Week -1]) by IV or SC injection once monthly for a total of 32 weeks. Doses were adjusted, if required, based on Hb level.
  This arm includes participants enrolled at CMUH.
- Mircera - KMUH: Participants received Mircera 80, 120, 200, or 360 mcg (based on the weekly dose of ESA participant received in the week preceding the switch to Mircera [Week -1]) by IV or SC injection once monthly for a total of 32 weeks. Doses were adjusted, if required, based on Hb level.
  This arm includes participants enrolled at KMUH.
- Mircera - BTCH: Participants received Mircera 80, 120, 200, or 360 mcg (based on the weekly dose of ESA participant received in the week preceding the switch to Mircera [Week -1]) by IV or SC injection once monthly for a total of 32 weeks. Doses were adjusted, if required, based on Hb level.
  This arm includes participants enrolled at BTCH.
Arm/Group | Mircera - CMUH | Mircera - KMUH | Mircera - BTCH | Mircera
Number analyzed (Participants) | 35 | 26 | 22 | 83
g/dL
  Baseline (n=35,26,22,83) | 10.7 (0.6) | 11.1 (0.6) | 10.8 (0.4) | 10.8 (0.6)
  Month 1 (n=35,26,22,83) | 10.7 (1.2) | 11.3 (0.8) | 10.9 (1.0) | 10.9 (1.0)
  Month 2 (n=34,26,21,81) | 10.8 (1.4) | 10.9 (1.1) | 11.2 (1.2) | 10.9 (1.3)
  Month 3 (n=33,22,20,75) | 10.8 (1.2) | 10.9 (1.0) | 11.8 (1.0) | 11.1 (1.1)
  Month 4 (n=31,22,19,72) | 10.9 (1.3) | 10.5 (1.3) | 11.4 (0.9) | 10.9 (1.3)
  Month 5 (n=28,21,19,68) | 11.0 (1.1) | 10.5 (1.2) | 11.5 (0.9) | 11.0 (1.1)
  Month 6 (n=28,20,19,67) | 10.9 (1.0) | 10.4 (1.2) | 11.4 (0.9) | 10.9 (1.1)
  Month 7 (n=27,20,19,66) | 11.3 (0.9) | 10.9 (1.5) | 11.0 (0.9) | 11.1 (1.1)
  Month 8 (n=26,19,19,64) | 11.5 (1.0) | 10.8 (0.9) | 11.1 (1.0) | 11.2 (1.0)

3. Secondary Outcome: Change in Hb Concentration Between Reference and Treatment Period
Description: as for outcome 2
Time Frame: Baseline, Months 1, 2, 3, 4, 5, 6, 7, 8
Population: ITT Population. Here, n signifies participants evaluable at specified time-point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera - CMUH | Mircera - KMUH | Mircera - BTCH | Mircera
Number analyzed (Participants) | 35 | 26 | 22 | 83
g/dL
  Change at Month 1 (n=35,26,22,83) | -0.0 (1.0) | 0.1 (0.8) | 0.1 (1.0) | 0.1 (0.9)
  Change at Month 2 (n=34,26,21,81) | 0.1 (1.3) | -0.3 (1.1) | 0.4 (1.3) | 0.0 (1.3)
  Change at Month 3 (n=33,22,20,75) | 0.2 (1.1) | -0.3 (1.2) | 1.0 (1.1) | 0.2 (1.2)
  Change at Month 4 (n=31,22,19,72) | 0.2 (1.4) | -0.7 (1.4) | 0.6 (1.1) | 0.0 (1.4)
  Change at Month 5 (n=28,21,19,68) | 0.4 (1.1) | -0.7 (1.2) | 0.7 (1.0) | 0.1 (1.3)
  Change at Month 6 (n=28,20,19,67) | 0.3 (1.2) | -0.8 (1.2) | 0.6 (1.0) | 0.0 (1.3)
  Change at Month 7 (n=27,20,19,66) | 0.7 (1.2) | -0.4 (1.6) | 0.2 (1.0) | 0.2 (1.3)
  Change at Month 8 (n=26,19,19,64) | 0.9 (1.3) | -0.4 (0.9) | 0.4 (1.2) | 0.4 (1.3)
Statistical Analysis 1: Comparison: Mircera - CMUH; Change from baseline to Month 1: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.9825, Paired t-test
Statistical Analysis 2: Comparison: Mircera - KMUH; Change from baseline to Month 1: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.5737, Paired t-test
Statistical Analysis 3: Comparison: Mircera - BTCH; Change from baseline to Month 1: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.5703, Paired t-test
Statistical Analysis 4: Comparison: Mircera; Change from baseline to Month 1: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.5684, Paired t-test
Statistical Analysis 5: Comparison: Mircera - CMUH; Change from baseline to Month 2: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.8235, Paired t-test
Statistical Analysis 6: Comparison: Mircera - KMUH; Change from baseline to Month 2: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.2384, Paired t-test
Statistical Analysis 7: Comparison: Mircera - BTCH; Change from baseline to Month 2: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.1634, Paired t-test
Statistical Analysis 8: Comparison: Mircera; Change from baseline to Month 2: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.7816, Paired t-test
Statistical Analysis 9: Comparison: Mircera - CMUH; Change from baseline to Month 3: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.3917, Paired t-test
Statistical Analysis 10: Comparison: Mircera - KMUH; Change from baseline to Month 3: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.1749, Paired t-test
Statistical Analysis 11: Comparison: Mircera - BTCH; Change from baseline to Month 3: analysis was performed using paired t-test; Test type: Superiority or Other; p < 0.001, Paired t-test
Statistical Analysis 12: Comparison: Mircera; Change from baseline to Month 3: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0905, Paired t-test
Statistical Analysis 13: Comparison: Mircera - CMUH; Change from baseline to Month 4: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.3766, Paired t-test
Statistical Analysis 14: Comparison: Mircera - KMUH; Change from baseline to Month 4: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0253, Paired t-test
Statistical Analysis 15: Comparison: Mircera - BTCH; Change from baseline to Month 4: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0209, Paired t-test
Statistical Analysis 16: Comparison: Mircera; Change from baseline to Month 4: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.8206, Paired t-test
Statistical Analysis 17: Comparison: Mircera - CMUH; Change from baseline to Month 5: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0907, Paired t-test
Statistical Analysis 18: Comparison: Mircera - KMUH; Change from baseline to Month 5: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0177, Paired t-test
Statistical Analysis 19: Comparison: Mircera - BTCH; Change from baseline to Month 5: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0050, Paired t-test
Statistical Analysis 20: Comparison: Mircera; Change from baseline to Month 5: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.3724, Paired t-test
Statistical Analysis 21: Comparison: Mircera - CMUH; Change from baseline to Month 6: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.2796, Paired t-test
Statistical Analysis 22: Comparison: Mircera - KMUH; Change from baseline to Month 6: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0066, Paired t-test
Statistical Analysis 23: Comparison: Mircera - BTCH; Change from baseline to Month 6: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0081, Paired t-test
Statistical Analysis 24: Comparison: Mircera; Change from baseline to Month 6: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.7853, Paired t-test
Statistical Analysis 25: Comparison: Mircera - CMUH; Change from baseline to Month 7: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0039, Paired t-test
Statistical Analysis 26: Comparison: Mircera - KMUH; Change from baseline to Month 7: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.3057, Paired t-test
Statistical Analysis 27: Comparison: Mircera - BTCH; Change from baseline to Month 7: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.3374, Paired t-test
Statistical Analysis 28: Comparison: Mircera; Change from baseline to Month 7: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.1410, Paired t-test
Statistical Analysis 29: Comparison: Mircera - CMUH; Change from baseline to Month 8: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0017, Paired t-test
Statistical Analysis 30: Comparison: Mircera - KMUH; Change from baseline to Month 8: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0677, Paired t-test
Statistical Analysis 31: Comparison: Mircera - BTCH; Change from baseline to Month 8: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.1608, Paired t-test
Statistical Analysis 32: Comparison: Mircera; Change from baseline to Month 8: analysis was performed using paired t-test; Test type: Superiority or Other; p = 0.0196, Paired t-test

4. Secondary Outcome: Mean Time Participants Spent Having Hb Concentration Within Target Range
Description: Target Hb concentration was between 10.0 and 12.0 g/dL.
Time Frame: Weeks 1 to 32
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mircera - CMUH | Mircera - KMUH | Mircera - BTCH | Mircera
Number analyzed (Participants) | 35 | 26 | 22 | 83
days | 112.6 (75.6) | 105.0 (74.0) | 107.6 (56.7) | 108.9 (69.8)

5. Secondary Outcome: Percentage of Participants Requiring Dose Adjustments
Description: Dose adjustment included: Dose Increase; No Change; and Dose Decreased. Participants who did not have this data available are reported as Not Done. Results are reported for overall treatment arm.
Time Frame: Baseline to Month 1; Month 1 to 2; Month 2 to 3; Month 3 to 4; Month 4 to 5; Month 5 to 6; Month 6 to 7; Month 7 to 8
Population: ITT population. Here, number of participants analyzed signifies participants who were evaluable for this outcome and n signifies participants who were evaluable for specified time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera
Number analyzed (Participants) | 81
percentage of participants
  Baseline to Month 1: Increase (n=81) | 7.4
  Baseline to Month 1: No Change (n=81) | 61.7
  Baseline to Month 1: Decrease (n=81) | 21.0
  Baseline to Month 1: Not Done (n=81) | 9.9
  Month 1 to Month 2: Increase (n=75) | 4.0
  Month 1 to Month 2: No Change (n=75) | 69.3
  Month 1 to Month 2: Decrease (n=75) | 16.0
  Month 1 to Month 2: Not Done (n=75) | 10.7
  Months 2 to 3: Increase (n=72) | 6.9
  Months 2 to 3: No Change (n=72) | 59.7
  Months 2 to 3: Decrease (n=72) | 19.4
  Months 2 to 3: Not Done (n=72) | 13.9
  Months 3 to 4: Increase (n=68) | 4.4
  Months 3 to 4: No Change (n=68) | 64.7
  Months 3 to 4: Decrease (n=68) | 16.2
  Months 3 to 4: Not Done (n=68) | 14.7
  Months 4 to 5: Increase (n=67) | 11.9
  Months 4 to 5: No Change (n=67) | 61.2
  Months 4 to 5: Decrease (n=67) | 11.9
  Months 4 to 5: Not Done (n=67) | 14.9
  Months 5 to 6: Increase (n=66) | 6.1
  Months 5 to 6: No Change (n=66) | 59.1
  Months 5 to 6: Decrease (n=66) | 21.2
  Months 5 to 6: Not Done (n=66) | 13.6
  Months 6 to 7: Increase (n=64) | 12.5
  Months 6 to 7: No Change (n=64) | 65.6
  Months 6 to 7: Decrease (n=64) | 9.4
  Months 6 to 7: Not Done (n=64) | 12.5
  Months 7 to 8: Increase (n=64) | 3.1
  Months 7 to 8: No Change (n=64) | 84.4
  Months 7 to 8: Decrease (n=64) | 0.0
  Months 7 to 8: Not Done (n=64) | 12.5

ADVERSE EVENTS:
Time Frame: 8 months
Description: Safety population included all enrolled participants. Adverse events are reported for overall treatment arm.
Arm/Group | Mircera
Serious Adverse Events (participants affected / at risk) | 14/86
Other Adverse Events (participants affected / at risk) | 79/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=86)
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Alcoholic liver disease (Hepatobiliary disorders) | 1
Chronic hepatitis (Hepatobiliary disorders) | 1
Abdominal infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Septic embolus (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 1
Labile blood pressure (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=86)
Hyperparathyroidism (Endocrine disorders) | 8
Abdominal distension (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 11
Regurgitation (Gastrointestinal disorders) | 6
Oedema peripheral (General disorders) | 12
Pyrexia (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 23
Urinary tract infection (Infections and infestations) | 7
Contusion (Injury, poisoning and procedural complications) | 5
Haemodialysis complication (Injury, poisoning and procedural complications) | 7
Procedural hypertension (Injury, poisoning and procedural complications) | 5
Procedural hypotension (Injury, poisoning and procedural complications) | 12
Wound (Injury, poisoning and procedural complications) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 13
Hyperphosphataemia (Metabolism and nutrition disorders) | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 10
Headache (Nervous system disorders) | 14
Insomnia (Psychiatric disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 24
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11
Dermatitis (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 14
Hypertension (Vascular disorders) | 28
Hypotension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.